CLINICAL TRIAL: NCT03989193
Title: Evaluation of Marginal Bone Loss Using Computer Guided Ridge Splitting With Simultaneous Implant Placement Versus Conventional Technique (a Randomized Clinical Trial)
Brief Title: Evaluation of Marginal Bone Loss Using Computer Guided Ridge Splitting Technique With Simultaneous Implant Placement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basel mohammed hamzah, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: guidedsplit surgerymsc
Record Dates: First submitted 2019-06-09; First posted 2019-06-18 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Marginal Bone Loss; Computer Guided; Ridge Splitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer guided alveolar ridge splitting technique (Experimental): Computer guided alveolar ridge splitting using piezo electric device and a 3D printed surgical guide. An L shaped splitting pattern with one crestal and one distal cut will be performed.
  Interventions: Device: Computer guided alveolar ridge splitting technique

INTERVENTIONS:
Device: Computer guided alveolar ridge splitting technique — The bone splitting technique could be performed using the piezoelectric system, calibrating the device on D1 setting and using profuse saline irrigation. The preparation sequence begins with CS3 insert until a total depth of 10mm was achieved across the entire extension of the ridge. The procedure continued with the CS1 insert and finally the CS2 insert.
  The vertical bone cuts through the cortical layer: At the distal end of the horizontal split, a vertical cut will made with the high-speed bur within the vicinity of the buccal plate to start the separation, with a full vertical depth of 13 mm. Final design of the splitting cut was L-shaped split. At the distal and the mesial end of the horizontal split, a vertical cut was made with the high-speed bur for a full vertical depth of 13mm.

SUMMARY:
This clinical report describes a technique for ridge splitting, and gradual expansion in the maxilla with simultaneous implant placement with in the split ridge, with the preservation of the thin buccal plate of bone for proper blood supply.

DETAILED DESCRIPTION:
All the procedures will perform under local anesthesia (mepivacain with levonordefrin). Horizontal Atrophic maxillary sectors will use for the development of the treatment sequence. All the patients will prepare initially with study models that permitted surgical and prosthetic planning as well as the non-strict surgical guide for intraoperative use. After application of conventional local anesthesia techniques, a full thickness incision 3 line pyramidal flap will be expose the defect ridge. The incision will extend to the next tooth or at least 5 mm more posterior from the end of the osteotomy indicated, securing direct observation of the alveolar crest.

With a direct view of the alveolar crest, if the ridge presented a width close to 1.5 mm, the ARST was performed immediately; if it presented less than 1.5 mm, then it was worn down with a diamond bur (low speed motor at 1800 rpm) to reduce the height, obtaining an improved alveolar crest width up to approximately 1.5 mm.

With this condition the bone splitting technique could be performed using the piezoelectric system (Piezotome2¨, Satelec Action, France), calibrating the device on the D1 setting and using profuse saline irrigation. The preparation sequence was begun with the CS3 insert until a total depth of 10 mm was achieved across the entire extension of the ridge. The procedure continued with the CS1 insert and finally the CS2 insert. The CS% insert was used in two patients with the possibility of widening the osteotomy segment; this sequence always achieved a complete extension in depth of application.

In the study group the vertical bone cuts through the cortical layer.

* At the distal end of the horizontal split: a vertical cut was made with the high-speed bur within the vicinity of the buccal plate of bone; for the start of the separation. With a full vertical depth of 13 mm. Final design of the splitting cut was (L-SHAPE) SPLIT The control group the vertical bone cuts through the cortical layer.
* At the distal and mesial end of the horizontal split: a vertical cut was made with the high-speed bur within the vicinity of the buccal plate of bone; for the start of the separation. With a full vertical depth of 13 mm corresponding and joining the previous vertical cut.

Using the expander to do the implants bed.-Preparation of the implant bed in the mesial end of the horizontal split using the spreading kit.-The final size spreader in the first implant osteotomy site with the first spreader in the second implant bed 3 mm apart. Dental implant placement. Placing the first implant in place while the separation kept preserved .placing the last spreader in the second implant osteotomy site. Bone deficiency is addressed by filling with osteoplastic material; a bio resorbing barrier membrane is arranged.

CBCT assessment For the calculation of marginal bone loss(MBL), the implant will use as a reference by adjusting the cross-sectional long axis in the center of the implant and bisecting it (showing the buccolingual and mesiodistal dimensions). On the cross-sectional view, a line will draw just parallel to the implant, starting at the crest of the labial plate of bone and ending at the apical level of the implant; height will recorded in millimeters. The same process was repeated from the palatal direction. The panoramic view (longitudinal cut) will utilized to calculate the mesial and distal bone heights in millimeters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thin maxillary ridge of 3 to 5 mm thickness of crestal alveolar bone (horizontal deficiency).
* Patients with free medical history and adequate proper oral hygiene.
* Patients of adequate alveolar bone height.
* Both genders males and females will be included.

Exclusion Criteria:

* General contraindications to implant surgery.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Lack of opposite occluding dentition/prosthesis in the area intended for implant placement.
* Active infection or severe inflammation in the area intended for implant placement.
* Need of bone augmentation procedures at implant placement.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* any 'complex case' if implants had to be placed in the aesthetic zone defined as second to second maxillary premolars.
* Patients participating in other studies, if the present protocol could not be properly followed.
* Requiring only single implant-supported crowns.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
the amount of marginal bone loss | 6 months
  the amount of marginal bone loss of thin narrow ridge after 6 months of splitting bone taking the implant as guide measured in mm determined on cone beam CT (panoramic and cross-sectional views).